CLINICAL TRIAL: NCT06349304
Title: Impact of Regular Consumption of Grape on Eye Health and Regulation of Advanced Glycation End-products in Singapore Older Adults
Brief Title: Impact of Grape Powder Consumption on Eye Health and Glycemic Status in Singapore Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S25
Record Dates: First submitted 2024-03-14; First posted 2024-04-05 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-04

CONDITIONS: Macula; Degeneration; Aging; Advanced Glycation End Products
Keywords: Vitis vinifera; Older adults; Inflammation; Glycemic status; Oxidative stress; Eye health
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Freeze-dried table grape powder (Experimental): Subjects in this group will be given pouches, each containing 46 g of freeze-dried table grape powder, with an instruction sheet on how to prepare the powder into a drink for consumption.They will consume one pouch a day.
  Interventions: Dietary Supplement: Freeze-dried table grape powder
- Placebo table grape powder (Placebo Comparator): Subjects in this group will be given pouches, each containing 46 g of placebo grape powder, with an instruction sheet on how to prepare the powder into a drink for consumption.They will consume one pouch a day.
  Interventions: Dietary Supplement: Placebo grape powder

INTERVENTIONS:
Dietary Supplement: Freeze-dried table grape powder — Consumption of grape powder as part of daily diet
  Arms: Freeze-dried table grape powder
Dietary Supplement: Placebo grape powder — Consumption of placebo grape powder as part of daily diet
  Arms: Placebo table grape powder

SUMMARY:
The purpose of this study is to understand the impacts of regular consumption of freeze-dried table grape powder on eye health and regulation of advanced glycation end products in Singapore older adults. The investigators hypothesize that regular consumption of freeze-dried table grape powder will promote improvements in eye health and lower levels of advanced glycation end products when compared to the placebo group.

DETAILED DESCRIPTION:
The study will be a 16-week, double-blind, randomized, placebo-controlled trial using a parallel study design. 46 adults (aged 60 - 85) will be recruited and randomly assigned to the intervention or placebo group to investigate whether regular consumption of freeze-dried table grape powder (46g/d) can improve eye health parameters, blood/skin AGE and glycemic status, and reduce inflammation and oxidative stress. This study will consist of 1 screening visit and 5 study visits with 4-week intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, aged between 60 and 85 years old inclusive
2. English-literate and able to give informed consent in English

Exclusion Criteria:

1. Smokers
2. Allergy to grapes or food dyes/additives, or had serious food allergies in the past
3. Known eye diseases (macular degeneration, cataracts, retinopathy or glaucoma), blindness in at least one eye or have had eye surgery
4. Unable to view bright lights or flashing lights
5. Has Type 1 or 2 diabetes, uremia, cardiovascular disease, abnormal kidney and liver function
6. Taking eye medication and/or dietary supplements for the eyes for the past 3 month
7. Taking supplements containing carotenoids (e.g. Vitamin A, lutein, zeaxanthin) for past 3 months
8. Currently on a specialised diet (e.g. vegetarian, vegan, weight loss diet, low fat diet
9. Consumes more than 2 alcoholic drinks per day i.e. one drink is defined as either 150ml of wine,340ml of beer/cider or 45ml of distilled spirit
10. Significant change in weight (≥ 3 kg body weight) in the past 3 months
11. Significant exercise pattern over the past 3 months defined as high-intensity exercise of more than 3 hours per week
12. Currently on anti-hypertensive, cholesterol-lowering or psychoactive drugs
13. Scored ≤ 7 on the abbreviated mental test
14. Poor peripheral venous access based on past experiences with blood draw
15. Participating in another clinical study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Macular pigment optical density | Week 0, Week 4, Week 8, Week 12, Week 16
  A measurement of macular pigment of the eye using a heterochromatic flicker photometry device. The measurements are in arbitrary units.
Visual acuity | Week 0, Week 4, Week 8, Week 12, Week 16
  Participants will read out letters on a ETDRS LogMAR chart at a fixed distance where letters becomes smaller as it goes down the chart. Tests results will be recorded in number of letters read, where the more letters the better the outcome.
Photostress recovery time | Week 0, Week 4, Week 8, Week 12, Week 16
  An ophthalmoscope will be used to shine a light into the participants eye for 10 seconds, and participants will be required to read letters off a chart the moment their vision returns to normal. The faster the recovery time, the better the outcome. Units will be in seconds
Visual function questionnaire 25 | Week 0, Week 4, Week 8, Week 12, Week 16
  A questionnaire to for participants to self-evaluate their perception of their current eye health based on general vision, ocular pain, near activities, distance activities, vision specific functions, driving, color vision and peripheral vision. The best possible score is 100 and worst possible score is 0.
Skin advanced glycation end products levels | Week 0, Week 4, Week 8, Week 12, Week 16
  Measurement of skin advanced glycation end products level using a skin autofluorescence device, where participants wlll be instructed to place their forearm over the device and a light will be shone and a reading can be captured by detecting fluorescence. The results will be presented as arbitrary units.
Dietary advanced glycation end products level | Week 0, Week 4, Week 8, Week 12, Week 16
  Participants will be instructed to record down 3-day food records, from Thursday to Saturday, before each clinical visit. This will be used to estimate their advanced glycation end products intake from food by referring to existing nutrient databases. Units will be based on a common advanced glycation end product measured, carboxymethyllysine (CML), thus the unit will be mg CML/ kg food
Blood advanced glycation end products levels | Week 0, Week 8 and Week 16
  Participants will have their blood drawn by medical professionals at the Occupational Health Clinic. The blood will be processed and stored. Measurements will be done using ultra-performance liquid chromatography coupled with mass spectrometry techniques to determine the levels of advanced glycation end products. Units will be in μg/mL.
Contrast sensitivity | Week 0, Week 4, Week 8, Week 12, Week 16
  Participants will read out letters on a ETDRS LogMAR chart at a fixed distance, where the letters differs in lightness to test participants' sensitivity to contrast. Tests results will be recorded in number of letters read, where the more letters the better the outcome.

SECONDARY OUTCOMES:
Concentration of tumour necrosis factor-α | Week 0, Week 8, Week 16
  The blood obtained from the participants will be processed for storage. Tumor necrosis factor-α results will be presented in ng/L according to the commercially available enzyme-linked immunosorbent assay kits.
Concentration of interleukin-6 | Week 0, Week 8, Week 16
  The blood obtained from the participants will be processed for storage. Interleukin-6 results will be presented in ng/L according to the commercially available enzyme-linked immunosorbent assay kits.
Concentration of high-sensitivity C-reactive protein | Week 0, Week 8, Week 16
  The blood obtained from the participants will be processed for storage. Analyses of inflammation markers include tumor necrosis factor-α, interleukin-6. high sensitivity C-reactive protein. Tumor necrosis factor-α and interleukin-6 results will be presented in ng/L according to the commercially available enzyme-linked immunosorbent assay kits. High-sensitivity C-reactive protein results will be obtained and presented in mg/L by commercial lab testing.
Concentration of fasting blood glucose | Week 0, Week 8, Week 16
  Fasting blood glucose will be measured using commercial lab testing using participants' blood, units will be in mmol/L.
Concentration of malondialdehyde | Week 0, Week 8, Week 16
  The blood obtained from the participants will be processed for storage. Analyses of malondialdehyde using commercially available enzyme-linked immunosorbent assay kits. Units for malondialdehyde will be in ng/L according to assay kit instructions.
Concentration of 8-isoprostaglandin-F2α | Week 0, Week 8, Week 16
  The blood obtained from the participants will be processed for storage. Analyses of 8-isoprostaglandin-F2α using commercially available enzyme-linked immunosorbent assay kits. Units for 8-isoprostaglandin-F2α will be in µmol/L according to assay kit instructions.
Skin carotenoid status | Week 0, Week 4, Week 8, Week 12, Week 16;
  Measured using a commercially available device that measured carotenoids using Raman spectroscopy. Results are in arbitrary units.
Concentration of insulin | Week 0, Week 8, Week 16
  Fasting blood insulin will be measured using commercial lab testing using participants' blood, units in μU/L.
Percentage of glycated hemoglobin | Week 0, Week 8, Week 16
  Glycated hemoglobin will be measured using commercial lab testing from participant's blood, units in percent.

OTHER OUTCOMES:
Measurement of height | Week 0, Week 4, Week 8, Week 12, Week 16
  Height will be measured using height-weight scale and units will be in cm.
Measurement of blood pressure | Week 0, Week 4, Week 8, Week 12, Week 16
  A blood pressure monitoring device available commercially will be used be to measure their systolic nad diastolic blood pressure.
Measurement of weight | Week 0, Week 4, Week 8, Week 12, Week 16
  Weight will be measured using height-weight scale and units will be in kg.
Measurement of waist circumference | Week 0, Week 4, Week 8, Week 12, Week 16
  Waist circumference will be measured using a measuring tape by a trained personnel, units in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, Ph.D., R.D., Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Faculty of Science, Department of Food Science and Technology, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept on NUS OneDrive with access limited only Dr Kim Jung Eun and her research staff. All data will be de-identified prior to statistical analyses.

REFERENCES:
- [Background] Hu W, Zheng R, Feng Y, Tan D, Chan Chung-Tsing G, Su X, Kim JE. Impacts of regular consumption of grapes on macular pigment accumulation in Singapore older adults: a randomized controlled trial. Food Funct. 2023 Sep 19;14(18):8321-8330. doi: 10.1039/d3fo02105j. PMID 37605542